CLINICAL TRIAL: NCT04338971
Title: Ipsihand Device Use in Stroke Patients to Assess Motor Recovery of the Upper Extremity and Functional Outcomes
Brief Title: Ipsihand Device Use in Stroke Patients to Assess Functional Motor Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ipsihand Use in Chronic Stroke
Record Dates: First submitted 2017-05-30; First posted 2020-04-08 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Stroke
Keywords: Rehabilitation; Brain-Computer Interface
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IpsiHand Device (Experimental): All participants will receive treatment with the IpsiHand Device.
  Interventions: Device: IpsiHand Therapy

INTERVENTIONS:
Device: IpsiHand Therapy — The IpsiHand system utilizes a Brain-Computer Interface (BCI) to enable operation of a robotic hand exoskeleton worn on the hand and wrist as participants are guided through a rehabilitation program on a tablet. Participants will complete 12 weeks of hometherapy with the IpsiHand system. Motor function of their impaired upper extremity will be evaluated at baseline, at 4-week intervals, and 12 weeks completion of IpsiHand use.

SUMMARY:
This study aims to evaluate the impact of the Neurolutions Upper Extremity Rehabilitation System, known as IpsiHand, on improving functional motor control for post-stroke patients with hemiparesis. The Neurolutions System is a brain-computer interface (BCI) comprised of a robotic orthosis, worn on the hand and wrist, and operated by the patient's brain waves which are measured by EEG electrodes. The system also utilizes a tablet interface to provide therapy instructions to the patient.

DETAILED DESCRIPTION:
Participants will complete 12 weeks of home therapy with the Neurolutions IpsiHand System. Outcomes will be based on a comparison of the patient's baseline measurements to post-therapy assessments.

ELIGIBILITY:
Inclusion Criteria:

* 6-months or more post stroke
* Presentation of upper extremity hemiparesis or hemiplegia
* Participants must english speaking
* Demonstrate intact cognition to provide informed consent
* Botox injections are allowed, and must continue regimen at regular intervals throughout the study

Exclusion Criteria -

* Not active in another clinical study
* Not receiving formal therapy for the upper extremity
* No use of other modalities or technologies to the upper extremity
* Cognitive Impairment: Short Blessed Test Score 9 or above
* Significant Spasticity: Modified Ashworth Scale score 3 or more at the elbow
* Significant Hemispatial Neglect: Mesulam Cancellation Test 3 or more unilaterally
* Insufficient Strength: Motricity Index score for shoulder abduction 18 - Any contractors of the affected upper extremity that would not allow the IpsiHand robotic exoskeleton to be worn comfortably and/or safely for device use

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Carter, MD, PhD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - Neurolutions, Santa Cruz, California
  - Neurolutions, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bundy DT, Souders L, Baranyai K, Leonard L, Schalk G, Coker R, Moran DW, Huskey T, Leuthardt EC. Contralesional Brain-Computer Interface Control of a Powered Exoskeleton for Motor Recovery in Chronic Stroke Survivors. Stroke. 2017 Jul;48(7):1908-1915. doi: 10.1161/STROKEAHA.116.016304. Epub 2017 May 26. PMID 28550098
- [Background] Cervera MA, Soekadar SR, Ushiba J, Millan JDR, Liu M, Birbaumer N, Garipelli G. Brain-computer interfaces for post-stroke motor rehabilitation: a meta-analysis. Ann Clin Transl Neurol. 2018 Mar 25;5(5):651-663. doi: 10.1002/acn3.544. eCollection 2018 May. PMID 29761128
- [Background] Zeiler SR, Krakauer JW. The interaction between training and plasticity in the poststroke brain. Curr Opin Neurol. 2013 Dec;26(6):609-16. doi: 10.1097/WCO.0000000000000025. PMID 24136129
- [Derived] Rustamov N, Souders L, Sheehan L, Carter A, Leuthardt EC. IpsiHand Brain-Computer Interface Therapy Induces Broad Upper Extremity Motor Rehabilitation in Chronic Stroke. Neurorehabil Neural Repair. 2025 Jan;39(1):74-86. doi: 10.1177/15459683241287731. Epub 2024 Sep 30. PMID 39345118

RESULTS

PARTICIPANT FLOW:
Groups:
- IpsiHand Intervention: This study was a prospective, non-randomized, self-controlled study performed in two phases at two investigational sites. 17 chronic stroke survivors (6 months or more post stroke) utilized the BCI Neurolutions IpsiHand System (the "device") at home for 12 weeks. During this time, data was collected at baseline, during, and upon completion of use of the Neurolutions IpsiHand System.
Period: Overall Study
Arm/Group | IpsiHand Intervention
Started | 24
Completed | 17
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- IpsiHand Intervention: This study was a prospective, non-randomized, self-controlled study performed in two phases at two investigational sites. 17 chronic stroke survivors (6 months or more post stroke) utilized the BCI Neurolutions IpsiHand System (the "device") at home for 12 weeks. During this time, data was collected at baseline, during, and upon completion of use of the Neurolutions IpsiHand System.
  IpsiHand is a device which includes a robotic exoskeleton that you wear on your forearm and hand, an EEG headset worn on your head, and a tablet which includes therapy software and guides you through daily therapy exercises.
  Once a participant completes an initial EEG screening, the participant completes a set of baseline measurements, the IpsiHand BCI device is then provided to the participants and are to be used a minimum of 5 days a week out of 7 days , for a total duration of 12 weeks. Participants are seen monthly throughout the 12-week duration while they are using the IpsiHand. After completion of device use, participants were asked to be evaluated 6 months after discontinuation of the IpsiHand to assess durability effects.
Arm/Group | IpsiHand Intervention
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Baseline Scores of the "Fugl Meyer Assessment of the Upper Extremity" Score [Mean (Standard Deviation); unit: score on a scale (range: 0 to 66 points)] — Mean average score on the "Fugl-Meyer Assessment of the Upper Extremity" assessment. This assessment has a total score on a scale range of 0 to 66 points. The lower the score, the lower motor function of the impaired upper extremity. The higher the score, the better motor function in the upper extremity. A score of 66 would indicate no motor impairments assessed in the upper extremity.
  score on a scale (range: 0 to 66 points) | 9.18 (5.836)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment - Upper Extremity
Description: The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The FMA is a score on a scale of 0 to 66 points. A lower score indicates impaired motor function in the upper extremity assessed. A higher score on the scale indicates better motor function of the upper extremity. A score of 66 would indicate there is no motor function impairment of the upper extremity.
Time Frame: "Fugl-Meyer Assessment - Upper Extremity" average change in points from the baseline average score and 12-week average score.
Measure: Mean (Standard Deviation); unit: point change for score on assessment
Groups:
- IpsiHand Intervention: Change in Fugl-Meyer Assessment of the Upper Extremity: This study was a prospective, non-randomized, self-controlled study performed in two phases at two investigational sites. 17 chronic stroke survivors (6 months or more post stroke) utilized the BCI Neurolutions IpsiHand System (the "device") at home for 12 weeks. During this time, data was collected at baseline, during, and upon completion of use of the Neurolutions IpsiHand System.
Arm/Group | IpsiHand Intervention: Change in Fugl-Meyer Assessment of the Upper Extremity
Number analyzed (Participants) | 17
point change for score on assessment | 9.18 (5.836)

2. Secondary Outcome: Arm Motor Ability Test Change Points on Scale From Baseline to 12 Weeks
Description: The Arm Motor Ability Test (AMAT is used to measure functional limitation in the upper extremity in rehabilitative trials enrolling individuals with stroke primarily. The measure requires clients to perform 28 common unilateral and bilateral UE tasks. Performance on each task is timed by the evaluator and rated by the evaluator using a 6-point Functional Ability Scale from 0 to 5. A score of 0 indicates no attempt moving the affected upper extremity in the task. A score of 5 indicates one is using their affected arm with full movement, normal. One can achieve a total a range of 0 points to 140 points
Time Frame: Change in AMAT score (points) from Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: change in points of score on a scale
Arm/Group | IpsiHand Intervention
Number analyzed (Participants) | 17
change in points of score on a scale | 12.65 (4.105)

ADVERSE EVENTS:
Time Frame: All adverse events were monitored throughout the study completion, an average of 2 years.
Arm/Group | IpsiHand Intervention
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04338971/Prot_SAP_001.pdf